CLINICAL TRIAL: NCT03964181
Title: Changing School Start Times: Impact on Student, Family, Teacher, and Community Health
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Lisa Meltzer, Associate Professor of Pediatrics, National Jewish Health
Other Study IDs: HS-3155; 75277 (Other Grant/Funding Number: Robert Wood Johnson Foundation Evidence for Action)
Record Dates: First submitted 2019-05-22; First posted 2019-05-28 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Sleep

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Students Grades 3-12
  Interventions: Other: Change in school start times
- Parents of Students Grades K-12
  Interventions: Other: Change in school start times
- School Based Teachers and Staff Grades K-12
  Interventions: Other: Change in school start times

INTERVENTIONS:
Other: Change in school start times — Elementary start times changed from 9:00 a.m. to 8:00 a.m.; middle school start times changed from 8:00 a.m. to 8:50 a.m.; high school start times changed from 7:10 a.m. to 8:20 a.m.

SUMMARY:
Sleep is not an optional luxury, but a fundamental biological need, essential for health and well-being. Insufficient sleep is a significant public health issue, with 69% of adolescents in America obtaining less than the minimum requirement of 8 hours of sleep per night. Early school start times has been identified as the most significant and modifiable factor that restricts sleep duration in adolescents. The American Academy of Pediatrics recommended in 2014 that all middle and high schools start no earlier than 8:30 a.m., yet few school districts have implemented this change. In fall 2017, the Cherry Creek School District, a diverse district of almost 55,000 students outside Denver, changed school start times. Although previous studies have shown increased sleep duration, decreased daytime sleepiness, and improved academics following start time changes for secondary students, there remains an urgent need to understand how this policy impacts health and well-being for all students, including youth in elementary school. Recognizing that students are part of a complex system that includes parents, school staff, and the community, this observational study will be a multi-year, broad-based evaluation that includes key stakeholders, multiple sources of quantitative data (i.e., surveys, academic records, district nursing electronic health records), contextual qualitative data (i.e., open-ended surveys and focus groups), and community-based outcomes (i.e., data on vehicle crashes and juvenile crimes). The primary hypothesis is that later school start times will have a positive impact on middle and high school students sleep and health outcomes, while earlier school start times will have a neutral impact on elementary school students sleep and health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Students in grades 3-12 enrolled in the school district
* Parents of students in grades K-12 enrolled in the school district
* School-based teachers and staff in grades K-12 in the school district

Exclusion Criteria:

* None

Min Age: 8 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants were drawn from the Cherry Creek School District outside of Denver, Colorado
Sampling Method: Non-Probability Sample
Enrollment: 118000 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in sleep duration from before start time change to 1 and 2 years after start time change | Typical bedtime and wake time, assessed prior to start time change, and 1 and 2 years after start time change
  Reported sleep from bedtime to wake time

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Meltzer LJ, McNally J, Plog AE, Siegfried SA. Engaging the community in the process of changing school start times: experience of the Cherry Creek School District. Sleep Health. 2017 Dec;3(6):472-478. doi: 10.1016/j.sleh.2017.08.005. Epub 2017 Oct 16. PMID 29157642
- [Result] Meltzer LJ, Wahlstrom KL, Plog AE, Strand MJ. Changing school start times: impact on sleep in primary and secondary school students. Sleep. 2021 Jul 9;44(7):zsab048. doi: 10.1093/sleep/zsab048. PMID 33855446
- [Result] Meltzer LJ, Wahlstrom KL, Plog AE, McNally J. Impact of changing school start times on parent sleep. Sleep Health. 2022 Feb;8(1):130-134. doi: 10.1016/j.sleh.2021.08.003. Epub 2021 Oct 9. PMID 34642123
- [Result] Meltzer LJ, Plog AE, Wahlstrom KL, Strand MJ. Biology vs. ecology: a longitudinal examination of sleep, development, and a change in school start times. Sleep Med. 2022 Feb;90:176-184. doi: 10.1016/j.sleep.2022.01.003. Epub 2022 Jan 10. PMID 35182977